CLINICAL TRIAL: NCT00936208
Title: To Evaluate the Safety, Efficacy, and Protection of Micardis 80 mg/Micardis Plus 80/12.5 mg From Cardiovascular Risks in a 24 Weeks Observational Study in Patients With Essential Hypertension Who Have at Least One Other Known Cardio-vascular Risk Factor
Brief Title: PRO-POWER: Hypertension With Risk Factors for a Duration of 24 Weeks With Micardis 80mg/Micardis Plus 80mg/12.5mg
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 502.584
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Results first posted 2012-07-02 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Essential hypertensive men and women

SUMMARY:
PRO-POWER is an observational cohort study for a period of 24 weeks. All recruited patients will have essential hypertension. In addition, the patients will have at least one other contributing risk factor for cardiovascular events. The study aims to evaluate the safety, efficacy and protection of Micardis 80mg/Micardis plus 80/12.5mg from cardiovascular risks in patients with essential hypertension

ELIGIBILITY:
Inclusion criteria:

* Male or female
* Aged 20 to 80 years old.
* adult with essential hypertension - either newly diagnosed and untreated, or previously treated and uncontrolled
* Sitting blood pressure: systolic BP > 140 mmHg but < 180 mmHg, and/or diastolic BP > 90 mmHg but < 110 mmHg)
* At least one cardiovascular known risk factor other than hypertension: diabetes/hyperglycaemia, cholesterol /dyslipidemia, a previous cardiovascular event, target organ damage, family history of hypertension or cardiovascular diseases, old age defined as > 55 years (Males), > 65 years (Females), smoking, overweight or obese patients or a combination of above risk factors
* Patients who are assessed to benefit from the intake of angiotensin II receptor blocker (ARB) monotherapy or as add-on medication

Exclusion criteria:

* Patients with contraindications to Telmisartan use (as per the Micardis® Tablets package insert).
* Known hypersensitivity to the active ingredient or to any of the excipients of Micardis® .
* Any other clinical condition which, in the opinion of the attending physician, would not allow safe administration of the study medications.
* Patients participating in any other clinical trial.
* Patients already on Micardis® alone or combination
* Pregnant females, or females breast feeding.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients in the Kingdom of Saudi Arabia, Egypt and United Arab Emirates
Sampling Method: Non-Probability Sample
Enrollment: 3184 (Actual)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (120):
- Egypt (30):
  - Boehringer Ingelheim Investigational Site 28, Al Fayyum
  - Boehringer Ingelheim Investigational Site 18, Alexandria
  - Boehringer Ingelheim Investigational Site 19, Alexandria
  - Boehringer Ingelheim Investigational Site 20, Alexandria
  - Boehringer Ingelheim Investigational Site 21, Alexandria
  - Boehringer Ingelheim Investigational Site 16, Alexandria West
  - Boehringer Ingelheim Investigational Site 17, Alexandria West
  - Boehringer Ingelheim Investigational Site 29, Asyut
  - Boehringer Ingelheim Investigational Site 10, Cairo
  - Boehringer Ingelheim Investigational Site 11, Cairo
  - Boehringer Ingelheim Investigational Site 12, Cairo
  - Boehringer Ingelheim Investigational Site 1, Cairo
  - Boehringer Ingelheim Investigational Site 2, Cairo
  - Boehringer Ingelheim Investigational Site 3, Cairo
  - Boehringer Ingelheim Investigational Site 4, Cairo
  - Boehringer Ingelheim Investigational Site 5, Cairo
  - Boehringer Ingelheim Investigational Site 6, Cairo
  - Boehringer Ingelheim Investigational Site 7, Cairo
  - Boehringer Ingelheim Investigational Site 8, Cairo
  - Boehringer Ingelheim Investigational Site 9, Cairo
  - Boehringer Ingelheim Investigational Site 22, Domiat
  - Boehringer Ingelheim Investigational Site 23, El Garbia
  - Boehringer Ingelheim Investigational Site 25, Fakous - El Sharkia
  - Boehringer Ingelheim Investigational Site 13, Kalioubya
  - Boehringer Ingelheim Investigational Site 27, Mansoura - El Dakahlia
  - Boehringer Ingelheim Investigational Site 30, Menofia
  - Boehringer Ingelheim Investigational Site 14, Minya
  - Boehringer Ingelheim Investigational Site 15, Minya
  - Boehringer Ingelheim Investigational Site 24, Poert Said
  - Boehringer Ingelheim Investigational Site 26, Zagazig - El Sharkia
- Saudi Arabia (71):
  - Boehringer Ingelheim Investigational Site 100, Eastern Region
  - Boehringer Ingelheim Investigational Site 101, Eastern Region
  - Boehringer Ingelheim Investigational Site 92, Eastern Region
  - Boehringer Ingelheim Investigational Site 93, Eastern Region
  - Boehringer Ingelheim Investigational Site 94, Eastern Region
  - Boehringer Ingelheim Investigational Site 95, Eastern Region
  - Boehringer Ingelheim Investigational Site 96, Eastern Region
  - Boehringer Ingelheim Investigational Site 97, Eastern Region
  - Boehringer Ingelheim Investigational Site 98, Eastern Region
  - Boehringer Ingelheim Investigational Site 99, Eastern Region
  - Boehringer Ingelheim Investigational Site 31, Riyadh
  - Boehringer Ingelheim Investigational Site 32, Riyadh
  - Boehringer Ingelheim Investigational Site 33, Riyadh
  - Boehringer Ingelheim Investigational Site 34, Riyadh
  - Boehringer Ingelheim Investigational Site 35, Riyadh
  - Boehringer Ingelheim Investigational Site 36, Riyadh
  - Boehringer Ingelheim Investigational Site 37, Riyadh
  - Boehringer Ingelheim Investigational Site 38, Riyadh
  - Boehringer Ingelheim Investigational Site 39, Riyadh
  - Boehringer Ingelheim Investigational Site 40, Riyadh
  - Boehringer Ingelheim Investigational Site 41, Riyadh
  - Boehringer Ingelheim Investigational Site 42, Riyadh
  - Boehringer Ingelheim Investigational Site 43, Riyadh
  - Boehringer Ingelheim Investigational Site 44, Riyadh
  - Boehringer Ingelheim Investigational Site 45, Riyadh
  - Boehringer Ingelheim Investigational Site 46, Riyadh
  - Boehringer Ingelheim Investigational Site 47, Riyadh
  - Boehringer Ingelheim Investigational Site 48, Riyadh
  - Boehringer Ingelheim Investigational Site 49, Riyadh
  - Boehringer Ingelheim Investigational Site 50, Riyadh
  - Boehringer Ingelheim Investigational Site 51, Riyadh
  - Boehringer Ingelheim Investigational Site 52, Riyadh
  - Boehringer Ingelheim Investigational Site 53, Riyadh
  - Boehringer Ingelheim Investigational Site 54, Riyadh
  - Boehringer Ingelheim Investigational Site 55, Riyadh
  - Boehringer Ingelheim Investigational Site 56, Riyadh
  - Boehringer Ingelheim Investigational Site 57, Riyadh
  - Boehringer Ingelheim Investigational Site 58, Riyadh
  - Boehringer Ingelheim Investigational Site 59, Western Region
  - Boehringer Ingelheim Investigational Site 60, Western Region
  - Boehringer Ingelheim Investigational Site 61, Western Region
  - Boehringer Ingelheim Investigational Site 62, Western Region
  - Boehringer Ingelheim Investigational Site 63, Western Region
  - Boehringer Ingelheim Investigational Site 64, Western Region
  - Boehringer Ingelheim Investigational Site 65, Western Region
  - Boehringer Ingelheim Investigational Site 66, Western Region
  - Boehringer Ingelheim Investigational Site 67, Western Region
  - Boehringer Ingelheim Investigational Site 68, Western Region
  - Boehringer Ingelheim Investigational Site 69, Western Region
  - Boehringer Ingelheim Investigational Site 70, Western Region
  - Boehringer Ingelheim Investigational Site 71, Western Region
  - Boehringer Ingelheim Investigational Site 72, Western Region
  - Boehringer Ingelheim Investigational Site 73, Western Region
  - Boehringer Ingelheim Investigational Site 74, Western Region
  - Boehringer Ingelheim Investigational Site 75, Western Region
  - Boehringer Ingelheim Investigational Site 76, Western Region
  - Boehringer Ingelheim Investigational Site 77, Western Region
  - Boehringer Ingelheim Investigational Site 78, Western Region
  - Boehringer Ingelheim Investigational Site 79, Western Region
  - Boehringer Ingelheim Investigational Site 80, Western Region
  - Boehringer Ingelheim Investigational Site 81, Western Region
  - Boehringer Ingelheim Investigational Site 82, Western Region
  - Boehringer Ingelheim Investigational Site 83, Western Region
  - Boehringer Ingelheim Investigational Site 84, Western Region
  - Boehringer Ingelheim Investigational Site 85, Western Region
  - Boehringer Ingelheim Investigational Site 86, Western Region
  - Boehringer Ingelheim Investigational Site 87, Western Region
  - Boehringer Ingelheim Investigational Site 88, Western Region
  - Boehringer Ingelheim Investigational Site 89, Western Region
  - Boehringer Ingelheim Investigational Site 90, Western Region
  - Boehringer Ingelheim Investigational Site 91, Western Region
- United Arab Emirates (19):
  - Boehringer Ingelheim Investigational Site 113, Abu Dhabi
  - Boehringer Ingelheim Investigational Site 114, Abu Dhabi
  - Boehringer Ingelheim Investigational Site 115, Abu Dhabi
  - Boehringer Ingelheim Investigational Site 116, Abu Dhabi
  - Boehringer Ingelheim Investigational Site 117, Abu Dhabi
  - Boehringer Ingelheim Investigational Site 118, Abu Dhabi
  - Boehringer Ingelheim Investigational Site 119, Abu Dhabi
  - Boehringer Ingelheim Investigational Site 120, Abu Dhabi
  - Boehringer Ingelheim Investigational Site 102, Dubai
  - Boehringer Ingelheim Investigational Site 103, Dubai
  - Boehringer Ingelheim Investigational Site 104, Dubai
  - Boehringer Ingelheim Investigational Site 105, Dubai
  - Boehringer Ingelheim Investigational Site 106, Dubai
  - Boehringer Ingelheim Investigational Site 107, Dubai
  - Boehringer Ingelheim Investigational Site 108, Dubai
  - Boehringer Ingelheim Investigational Site 109, Dubai
  - Boehringer Ingelheim Investigational Site 110, Dubai
  - Boehringer Ingelheim Investigational Site 111, Dubai
  - Boehringer Ingelheim Investigational Site 112, Sharjah city

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3184 patients were enrolled but treatment was unknown in 89 patients. Therefore, 3095 patients were analysed.
Groups:
- Micardis 80mg: One tablet of Micardis 80mg per day
- Micardis Plus 80mg / 12.5mg: One tablet of Micardis Plus 80 / 12.5mg per day
Period: Overall Study
Arm/Group | Micardis 80mg | Micardis Plus 80mg / 12.5mg
Started | 1499 | 1596
Completed | 1462 | 1574
Not Completed | 37 | 22
Not completed — Protocol Violation | 37 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Micardis 80mg | Micardis Plus 80mg / 12.5mg | Total
Number analyzed (Participants) | 1499 | 1596 | 3095
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was given for 1457 patients in the Micardis 80mg group and for 1569 patients in the Micardis Plus 80/12.5mg group.
  years | 49.8 (10.4) | 53.1 (9.8) | 51.5 (10.2)
Gender [Number; unit: participants] — Gender was given for 1431 patients in the Micardis 80mg group and for 1547 patients in the Micardis Plus 80/12.5mg group.
  participants
    Female | 500 | 434 | 934
    Male | 931 | 1113 | 2044
Framingham score at baseline [Mean (Standard Deviation); unit: Units on a scale] — The baseline Framingham score was given for 1349 patients in the Micardis 80mg group and for 1482 patients in the Micardis Plus 80/12.5mg group. The score represent the cardiovascular risk and ranges from 0 (no risk) to 100% (complete risk).
  Units on a scale | 15.7 (12.3) | 20.6 (12.5) | 18.6 (12.6)
International Renal Interest Society (IRIS) II score at baseline [Mean (Standard Deviation); unit: Units on a scale] — The baseline IRIS II score was given for 1122 patients in the Micardis 80mg group and for 1314 patients in the Micardis Plus 80/12.5mg group. The score represent the risk for vascular complication in type to diabetes mellitus and ranges from 0 (no risk) to 100% (complete risk).
  Units on a scale | 35.8 (33.8) | 37.1 (32.2) | 36.1 (32.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Diastolic Blood Pressure From Baseline at Week 24
Description: The change from baseline reflects the week 24 value minus the baseline value.
Time Frame: Baseline and Week 24
Population: Full Analysis Set (FAS): Patients with Blood Pressure data available at baseline and at week 24
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Micardis 80mg | Micardis Plus 80mg / 12.5mg
Number analyzed (Participants) | 1462 | 1574
mmHg | -15.3 (8.6) | -18.3 (8.4)

2. Primary Outcome: Change in Systolic Blood Pressure From Baseline at Week 24
Description: The change from baseline reflects the week 24 value minus the baseline value.
Time Frame: Baseline and Week 24
Population: Full Analysis Set (FAS): Patients with Blood Pressure data available at baseline and at week 24
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Micardis 80mg | Micardis Plus 80mg / 12.5mg
Number analyzed (Participants) | 1462 | 1574
mmHg | -26.6 (13.7) | -32.8 (15.0)

3. Secondary Outcome: Framingham Score at Week 24
Description: The Framingham score represent the cardiovascular risk and ranges from 0 (no risk) to 100% (complete risk).
Time Frame: Week 24
Population: Patients of Full Analysis Set (FAS) with values of the framingham score at baseline and at week 24
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Micardis 80mg | Micardis Plus 80mg / 12.5mg
Number analyzed (Participants) | 1349 | 1482
Units on a scale | 10.6 (8.4) | 14.2 (9.7)

4. Secondary Outcome: Change in the Framingham Score From Baseline at Week 24
Description: The change from baseline reflects the week 24 value minus the baseline value. The Framingham score represent the cardiovascular risk and ranges from 0 (no risk) to 100% (complete risk).
Time Frame: Baseline and Week 24
Population: Patients of Full Analysis Set (FAS) with values of the framingham score at baseline and at week 24
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Micardis 80mg | Micardis Plus 80mg / 12.5mg
Number analyzed (Participants) | 1349 | 1482
Units on a scale | -5.2 (8.7) | -6.3 (8.4)

5. Secondary Outcome: International Renal Interest Society (IRIS) II Score at Week 24
Description: The IRIS II score represent the risk for vascular complication in type to diabetes mellitus and ranges from 0 (no risk) to 100% (complete risk).
Time Frame: Week 24
Population: Patients of Full Analysis Set (FAS) with values of the IRIS II score at baseline and at week 24
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Micardis 80mg | Micardis Plus 80mg / 12.5mg
Number analyzed (Participants) | 1122 | 1314
Units on a scale | 30.9 (30.3) | 31.7 (28.8)

6. Secondary Outcome: Change in the IRIS II Score From Baseline at Week 24
Description: The change from baseline reflects the week 24 value minus the baseline value. The IRIS II score represent the risk for vascular complication in type to diabetes mellitus and ranges from 0 (no risk) to 100% (complete risk).
Time Frame: Baseline and Week 24
Population: Patients of Full Analysis Set (FAS) with values of the IRIS II score at baseline and at week 24
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Micardis 80mg | Micardis Plus 80mg / 12.5mg
Number analyzed (Participants) | 1122 | 1314
Units on a scale | -5.8 (13.9) | -7.0 (14.7)

7. Secondary Outcome: Change From Baseline in Urinary Microalbuminuria (Urine Dipstick Test Results)
Description: The change from baseline reflects the shift from baseline in urinary dipstick test results to week 24
Time Frame: Baseline and Week 24
Population: Patients of Full Analysis Set (FAS) with values of the dipstick test at baseline and at week 24
Measure: Number; unit: participants
Arm/Group | Micardis 80mg | Micardis Plus 80mg / 12.5mg
Number analyzed (Participants) | 1390 | 1514
participants
  Shift from baseline 0 to end-of-study 0 | 821 | 668
  Shift from baseline 0 to end-of-study 30 | 21 | 26
  Shift from baseline 0 to end-of-study 100 | 1 | 9
  Shift from baseline 0 to end-of-study 500 | 0 | 0
  Shift from baseline 30 to end-of-study 0 | 220 | 264
  Shift from baseline 30 to end-of-study 30 | 114 | 141
  Shift from baseline 30 to end-of-study 100 | 4 | 0
  Shift from baseline 30 to end-of-study 500 | 0 | 0
  Shift from baseline 100 to end-of-study 0 | 65 | 90
  Shift from baseline 100 to end-of-study 30 | 91 | 197
  Shift from baseline 100 to end-of-study 100 | 11 | 38
  Shift from baseline 100 to end-of-study 500 | 0 | 0
  Shift from baseline 500 to end-of-study 0 | 3 | 12
  Shift from baseline 500 to end-of-study 30 | 9 | 25
  Shift from baseline 500 to end-of-study 100 | 21 | 35
  Shift from baseline 500 to end-of-study 500 | 9 | 9

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Micardis 80mg | Micardis Plus 80mg / 12.5mg
Serious Adverse Events (participants affected / at risk) | 0/1499 | 0/1596
Other Adverse Events (participants affected / at risk) | 0/1499 | 0/1596

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.